CLINICAL TRIAL: NCT01124994
Title: Endomicroscopy-targeted Endoscopic Mucosa Resection for Barrett's Oesophagus-associated Neoplasia
Brief Title: Confocal Laser Endomicroscopy and Endoscopic Mucosal Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Werner Dolak, MD, Prinicpal Investigator, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EK 697/2009
Record Dates: First submitted 2010-05-17; First posted 2010-05-18 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Barrett's Mucosa With High Grade Intraepithelial Neoplasia (HGIEN)
Keywords: Barrett's oesophagus; High grade intraepithelial neoplasia (HGIEN)
MeSH Terms: conditions — Barrett Esophagus | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mucosectomy (Active Comparator): Patients in this arm are undergoing mucosctomy after previous confocal laser endomicroscopy.
  Interventions: Procedure: Endoscopic mucosal resection

INTERVENTIONS:
Procedure: Endoscopic mucosal resection — Confocal laser endomicroscopy will be used to target endoscopic mucosal resection of Barrett's oesophagus-associated neoplasia

SUMMARY:
The accurate detection and therapy of adenocarcinoma originating from Barrett's oesophagus is challenging as current endoscopic techniques are unreliable for both the detection of high grade intraepithelial neoplasia (HGIN) within Barrett's mucosa and the correct measurement of the dimension of such neoplastic lesions. Confocal laser endomicroscopy (CLE) is a promising technology that could help to close this gap. Relying on first clinical trials of CLE, which showed remarkable results for the detection of Barrett's associated neoplasia, the investigators want to use CLE as targeting tool for endoscopic mucosal resection of HGIN in patients suffering from Barrett's oesophagus. CLE-mapping of neoplastic lesions will be documented and compared to the later performed histological evaluation of the resected specimen. If CLE is passing our challenge this will be another valuable proof of its high potential as reliable new endoscopic technology. Its usage could increase the en-bloc resection rate and decrease the amount of repetitive resections, which would remarkably improve the patients comfort.

DETAILED DESCRIPTION:
Introduction

Barrett's oesophagus is a common complication in patients suffering from gastro-oesophageal reflux disease (GERD). By means of chronic acid exposure the squamous epithelium of the oesophagus turns into a specialised columnar epithelium (SCE) with goblet cells. This histological change is prevalent in 1% of the normal population, and in up to 4, 9% of patients with reflux symptoms [1]. Although the Barrett's epithelium itself does not necessarily cause additional symptoms, its presence has to be diagnosed accurately, since affected patients are at increased risk of 0.5% per year of developing Barrett's associated cancer. An important prognostic factor is made up by the grade of dysplasia within the Barrett's mucosa. While most patients with no dysplasia or low-grade dysplasia remain clinically inconspicuous, the annual risk of developing cancer is up to 10% in those patients with high-grade dysplasia. If a Barrett's associated neoplastic lesion is found during endoscopy, Barrett's associated cancer is also present at another site of Barrett's oesophagus in up to 30% [2].

Consequently, they undergo periodically screening, consisting of endoscopy of the oesophagus with 4-quadrant biopsy every 2 to 3 cm or, in case of HGIN, local ablative therapy. The time period between controls depends on the grade of dysplasia diagnosed at upper gastrointestinal endoscopy. If no dysplasia is present, the recommended follow-up period is less than 5 years. In case of low grade dysplasia endoscopic controls should be performed every year. Patients with high grade dysplasia should be examined every 3 months or prepared for a therapeutic intervention [3].

Early detection of Barrett's associated neoplasms, which can be histologically classified as adenocarcinoma, has important therapeutic implications. Cancerous infiltration of submucosal structures is associated with a significant risk of lymph node metastases and should be therefore treated by surgery. However, oesophagectomy has been shown to suffer from mortality rates between 3 and 12%, apart from substantial short- and long-term morbidity. Hence it is essential to detect early neoplastic lesions to have a broader range of therapeutic options at disposal. Patients with high grade intraepithelial neoplasia (HGIN) or mucosal cancer are perfect candidates for curative endoscopic interventions like endoscopic ablation (with radiofrequency, for example), endoscopic submucosal dissection (ESD) or endoscopic mucosal resection (EMR). The latter techniques are preferred as the resected specimens can be evaluated histologically, which provides definite information about the invasion depth and whether the resection borders are free from neoplastic tissue. Because of high rates of newly occurring neoplasia, remaining areas of Barrett's mucosa should be ablated or resected after histological confirmation of Barrett's oesophagus associated neoplasia [3, 4].

Trying to improve the diagnostic yield in the surveillance of patients with high risk for Barrett's oesophagus associated neoplasia, many new endoscopic inventions have been introduced into the management of Barrett's oesophagus in order to optimize the detection rates of early lesions. Among those are developments that improved the image quality of conventional white light endoscopes like high-resolution and high-definition endoscopes. Another approach, called chromoendoscopy, uses in vivo staining with methylene blue, indigo carmine or acetic acid. These dyes help to increase the tissue contrast which leads to improvement of detection rates comparable to high-resolution endoscopy. High contrast levels without staining agents can be achieved by the use of narrow band imaging (NBI). This technology additionally improves the visibility of capillaries, veins and other subtle tissue structures by the use of light with wavelength restricted to small bands in the blue and green spectrum. In a prospective randomized crossover study it showed equal results to high-resolution endoscopy plus indigo carmine [4, 5].

The newest development that has been introduced in the endoscopic management of the gastrointestinal tract is the so called confocal laser endomicroscope (CLE). Confocal microscopy was developed by Marvin Minsky in the late 1950s. Its principle is the microscopic scanning of focal points below the surface of an object. In comparison to conventional light microscopy it uses a special filter system to avoid image overlapping by surrounding tissue. In detail, a light source (normally a laser) is focused by a microscope objective lens to a diffraction limited spot on or inside the object. Light that is scattered, or fluorescence excited (achieved through fluorescein staining, for example) and emitted, at the focus in the sample will partially return back through the optics along the path from which it arrived. A beam-splitter placed into the path reflects the return light towards a detector. The optics will focus the light from the focal point in the specimen to its conjugate focus near the detector (hence the technology is termed "con-focal"). Here a spatial filter ("pinhole") is used to extinguish all light deriving from areas outside the focal point. Light reflections from the focal point itself will be forwarded to the detector which is connected to a computer system that digitalises the optical signal and creates the in vivo histological image [6].

Focussing on its clinical impact, confocal microscopy is the first technique to allow in vivo evaluation of tissue structures beneath their surface. Because of many breakthroughs in miniaturisation (mostly in the 1990s) this technology could be applied for intraluminal use in gastroenterology, integrated into a otherwise standard endoscope. It allows the in vivo histological visualisation of the upper 250 micrometers of all walls within the gastrointestinal tract, additionally to the normal function of white light endoscopy (provided by two separate screens on top of the workstation) [6].

Using CLE in a first clinical approach, Kiesslich et al. found high sensitivity and specificity rates for the detection of Barrett's oesophagus as well as for the prediction of Barrett's associated neoplastic changes - for both results CLE derived pictures were compared to conventional histology [7]. In a first prospective, randomized, double-blind, controlled, crossover trial Dunbar et al. proved these findings, as CLE-targeted biopsies had a higher diagnostic yield for Barrett's oesophagus associated neoplasia than standard endoscopy with 4-quadrant random biopsy [8].

Study Aims

In our clinical investigation we want to use confocal laser endomicroscopy (CLE) to accurately target Barrett's oesophagus associated neoplasia for subsequent endoscopic mucosal resection (EMR). To our knowledge this combination is only documented in one case report so far, describing the successful resection of a high-grade dysplastic Barrett-segment by the use of CLE-targeted EMR [9].

We want to show that CLE is suitable to detect the exact borders of high grade intraepithelial neoplasia. In our experience this feasibility cannot be reliably provided by any other established technique like chromoendoscopy or narrow band imaging, which often causes the need for re-treatment or even surgery.

To guarantee accurate documentation of mucosal CLE-mapping, the dimensions of the neoplastic lesion will be marked in terms of colour, photographed by simultaneously available white light endoscopy and finally evaluated by histological assessment of the specimen. Analysing the borders of the resected specimen in concern of tumour infiltration we will be able to calculate the en-bloc resection rate of CLE-targeted EMR.

In order to evaluate CLE concerning true negative results we will resect all remaining mucosal areas affected by Barrett within the second phase of the examination or (if the lesions are too big for one-time resection) within a second examination. Once again, CLE will be applied for all lesions to search for malignancies. If CLE detects further areas of neoplasia, CLE-mapping as mentioned above will be performed. All resected tissue parts will be evaluated histologically to check the results of CLE.

If CLE provides reliable data in our investigation this would be a big step on the way to establishing this new technology within the pre-interventional endoscopic management of patients suffering from Barrett's oesophagus. This could help to increase the en-bloc resection rate, decrease the amount of repetitive resections and consequentially improve the patients comfort.

Study Design

Prospective clinical trial without randomisation or blinding

Study Population

Patients referred to our department for endoscopic mucosal resection (EMR) of Barrett's mucosa with high grade intraepithelial neoplasia (HGIN) that has been detected during routine upper endoscopy or Barrett's surveillance endoscopy at our department or at another hospital.

Exclusion criteria:

* patients allergic to one of the drug components (including drugs used for conscious sedation like propofol or midazolam as well as fluorescein, the fluorescent dye used for CLE )
* patients presenting with contraindications to EMR (low platelet count, therapeutic anticoagulation, coagulation disorders)
* refusal to participate in the study

Methods

Our investigation will be performed at the Medical University of Vienna, department of medicine III, clinical division of gastroenterology and hepatology. Patient recruitment will start on the 1st of July 2010. The study will last for two years. The number of patients included within this period will be 40, based on the current number of EMR performed at our department for Barrett's with intraepithelial neoplasia.

All patients who fulfil the listed inclusion criteria, will receive the patient information form of this study together with the usual informed consent form of the respective endoscopic examination they are about to undergo. Patient information will be done at least 24 hrs. before the intervention, as practised at our unit. If the patient agrees to participate in the study he will be prepared for endoscopy with our confocal laser endomicroscope (Pentax EC3870K with the ISC-1000 confocal endomicroscopy processor - Pentax, Tokyo, Japan and Optiscan Pty Ltd, Notting Hill, Victoria, Australia) by administration of intravenous propofol and/or midazolam as routinely used for conscious sedation during endoscopic procedures at our department. Additionally, 5-10 ml of a 10% solution of fluorescein sodium will be administered intravenously to enhance tissue fluorescence during endomicroscopy.

All drugs will be administered by medical specialists (such as the project director), assistant doctors (such as the project assistant) or registered nurses, as routinely practised at our institution.

Ethical implications

Confocal laser endomicroscopy is a safe new technique that has already been studied in clinical trials [7, 8]. Its safety is being guaranteed by the use of low intensity laser light that can at worst cause local bleaching of fluorescein containing cells, which is harmless, reversible and even used as diagnostic sign in experimental conditions [6].

Endoscopic mucosal resection is a well established technique for the minimal invasive, non-surgical curative treatment of intramucosal neoplasia. It has been studied in many clinical trials and is routinely performed at our unit for lesions in the oesoophagus, the stomach, duodenum and colo-rectum. Although severe complications like prolonged bleeding or perforations can potentially occur, the risk/benefit profile of this procedure is very good, compared to surgical treatments of neoplastic diseases of the oesophagus [10].

This study protocol has been submitted to the ethic commission of the Medical University of Vienna (EK-Nr. 697/2009) and was handled at the meeting on the 8th of September 2009. A positive vote was already delivered to our institution in written form.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to our department for endoscopic mucosal resection (EMR) of Barrett's mucosa with high grade intraepithelial neoplasia (HGIN) that has been detected during routine upper endoscopy or Barrett's surveillance endoscopy at our department or at another hospital.

Exclusion Criteria:

* patients allergic to one of the drug components (including drugs used for conscious sedation like propofol or midazolam as well as fluorescein, the fluorescent dye used for CLE )
* patients presenting with contraindications to EMR (low platelet count, therapeutic anticoagulation, coagulation disorders)
* refusal to participate in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-07; Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Accuracy of CLE-EMR | 2 years
  Accuracy of CLE to detect the exact borders of high grade intraepithelial neoplasia within Barrett's epithelium, confirmed by histological evaluation of resected specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Puespoek, MD, Study Director — Medical University of Vienna; Werner Dolak, MD, Principal Investigator — Medical University of Vienna, Department of Internal Medicine III, Division of Gastroenterology and Hepatology
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Background] Holscher AH, Vallbohmer D, Bollschweiler E. Early Barrett's carcinoma of the esophagus. Ann Thorac Cardiovasc Surg. 2008 Dec;14(6):347-54. No abstract available. PMID 19131920
- [Background] Shaheen NJ, Richter JE. Barrett's oesophagus. Lancet. 2009 Mar 7;373(9666):850-61. doi: 10.1016/S0140-6736(09)60487-6. PMID 19269522
- [Background] Spechler SJ. Dysplasia in Barrett's esophagus: limitations of current management strategies. Am J Gastroenterol. 2005 Apr;100(4):927-35. doi: 10.1111/j.1572-0241.2005.41201.x. PMID 15784042
- [Background] Curvers WL, Bansal A, Sharma P, Bergman JJ. Endoscopic work-up of early Barrett's neoplasia. Endoscopy. 2008 Dec;40(12):1000-7. doi: 10.1055/s-0028-1103409. Epub 2008 Dec 8. No abstract available. PMID 19065483
- [Background] Kara MA, Peters FP, Rosmolen WD, Krishnadath KK, ten Kate FJ, Fockens P, Bergman JJ. High-resolution endoscopy plus chromoendoscopy or narrow-band imaging in Barrett's esophagus: a prospective randomized crossover study. Endoscopy. 2005 Oct;37(10):929-36. doi: 10.1055/s-2005-870433. PMID 16189764
- [Background] Kiesslich R, Galle P, Neurath M. Atlas of endomicroscopy. Springer Medical Publishing. 2008
- [Background] Kiesslich R, Gossner L, Goetz M, Dahlmann A, Vieth M, Stolte M, Hoffman A, Jung M, Nafe B, Galle PR, Neurath MF. In vivo histology of Barrett's esophagus and associated neoplasia by confocal laser endomicroscopy. Clin Gastroenterol Hepatol. 2006 Aug;4(8):979-87. doi: 10.1016/j.cgh.2006.05.010. Epub 2006 Jul 13. PMID 16843068
- [Background] Dunbar KB, Okolo P 3rd, Montgomery E, Canto MI. Confocal laser endomicroscopy in Barrett's esophagus and endoscopically inapparent Barrett's neoplasia: a prospective, randomized, double-blind, controlled, crossover trial. Gastrointest Endosc. 2009 Oct;70(4):645-54. doi: 10.1016/j.gie.2009.02.009. Epub 2009 Jun 25. PMID 19559419
- [Background] Leung KK, Maru D, Abraham S, Hofstetter WL, Mehran R, Anandasabapathy S. Optical EMR: confocal endomicroscopy-targeted EMR of focal high-grade dysplasia in Barrett's esophagus. Gastrointest Endosc. 2009 Jan;69(1):170-2. doi: 10.1016/j.gie.2008.03.1068. Epub 2008 Jun 25. No abstract available. PMID 18582880
- [Background] Ahmadi A, Draganov P. Endoscopic mucosal resection in the upper gastrointestinal tract. World J Gastroenterol. 2008 Apr 7;14(13):1984-9. doi: 10.3748/wjg.14.1984. PMID 18395896